CLINICAL TRIAL: NCT02178540
Title: A Multi-center, Human Factors Engineering (HFE) Usability Study in Cystic Fibrosis Patients to Validate the Approved Instructions for Use (IFU) of TOBI® Podhaler™ (Tobramycin Inhalation Powder) Using Placebo Capsules
Brief Title: Study to Validate the Instructions for Use of TOBI® Podhaler™ in Cystic Fibrosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CTBM100C2412
Record Dates: First submitted 2014-06-24; First posted 2014-06-30 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
Keywords: Human factors, TOBI® Podhaler™, Instructions For use, IFU, CF patients
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open label (Other): one dose (4 capsules) of placebo
  Interventions: Drug: Placebo; Device: Tobi Podhaler

INTERVENTIONS:
Drug: Placebo — one dose (4 capsules) of placebo
Device: Tobi Podhaler — The capsule containing the study medication has to be released from the blister card, be inserted into the Podhaler device, actuated and the study drug be inhaled according to instructions for use

SUMMARY:
The purpose of this actual use human factors (HF) study is to validate the approved US TOBI Podhaler Instructions for Use (IFU), by establishing that the IFU effectively communicates the information necessary to achieve safe and effective use of the Podhaler device.

DETAILED DESCRIPTION:
The objective of the HF study is to determine whether cystic fibrosis patients in the US, representative of potential TOBI Podhaler users, can understand and follow the approved IFU and the extent to which the approved IFU supports safe and effective use of the Podhaler device.

This study is an 'actual use' study, in that patients will inhale the contents of placebo capsules through the Podhaler device.

Due to the use of placebo capsules, the study is considered a clinical study and will be conducted accordingly. The study is therefore a human factors observational use study conducted within a clinical study. It is an open label, unblinded, non-randomized study and consists of two visits. At visit 2 patients who are eligible will participate in a human factor assessment to determine whether or not a patient understands the IFU content and can demonstrate safe and effective use of the Podhaler device.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 6 years and older at screening
* Confirmed diagnosis of CF
* Pulmonary function FEV1 value at least 25% of normal predicted values
* Must be physically and cognitively able to read, alone or with the assistance of their caregiver

Exclusion Criteria:

* Subjects currently enrolled in studies that are not considered observational noninvestigational studies.
* Subjects who have used the Podhaler device previously
* Hemoptysis more than 60mL at any time within 30 days prior to study drug administration
* History of hypersensitivity to inhaled dry powder
* Signs and symptoms of acute pulmonary disease, e.g., pneumonia, pneumothorax

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (12):
- United States (12):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Long Beach, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Ventura, California
  - Novartis Investigative Site, Washington D.C., District of Columbia
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label: one dose (4 capsules) of matching placebo to Tobramycin inhalation powder hard capsule
Period: Overall Study
Arm/Group | Open Label
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.9 (7.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: The Use of the Approved US TOBI Podhaler Instructions for Use (IFU) to Communicates the Information Necessary to Achieve Safe and Effective Use of the Podhaler Device
Description: Recording all use errors and close calls associated with inhalation of one dose of TOBI Podhaler (i.e., inhaling the contents of four placebo capsules via the Podhaler device) by subjects (CF patients, and caregivers, if applicable). The study population consisted of CF patients (and caregivers) naïve to the Podhaler device and untrained in the use of the device. Assessing the root cause of use errors and close calls for 6 defined critical errors (agreed with the FDA) and establishing those which can be attributed to a lack of clarity or presence of ambiguities in the IFU content, i.e., errors attributable to a failure to understand the IFU.
Time Frame: 1 Day
Population: The Full Analysis Set (FAS) included all enrolled patients who completed an HF assessment as defined by completion of inhalation of the contents of at least one capsule and related HF assessment.
Measure: Number; unit: Patients failing to understand IFU
Arm/Group | Open Label
Number analyzed (Participants) | 45
Patients failing to understand IFU
  Failure to open blisters | 0
  Attempting to swallow the capsule | 0
  Placing capsule into the mouthpiece | 0
  Failure to pierce any of the 4 capsules (caps)* | 3
  Failure to inhale from all 4 capsules | 0
  Failure to inhale all powder from any of 4 caps† | 6

ADVERSE EVENTS:
Groups:
- Open Label (6-10) Years Old: one dose (4 capsules) of matching placebo to Tobramycin inhalation powder hard capsule
Arm/Group | Open Label (6-10) Years Old | Total - All Participants | Open Label (11-17)Years Old | Open Label (>=18) Years Old
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/45 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/45 | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label (6-10) Years Old (N=15) | Total - All Participants (N=45) | Open Label (11-17)Years Old (N=15) | Open Label (>=18) Years Old (N=15)
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Pulmonary function test decreased (Investigations) | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Participating patients were naïve to the Podhaler device, and untrained in its use. Patients accessed only the approved IFU document. Open label study using placebo only, potentially impacting perception of need to complete tasks fully.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial